CLINICAL TRIAL: NCT04573283
Title: A Prospective Cohort Study of Metabolic Associated Fatty Liver Disease in China
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-201506
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Associated Fatty Liver Disease
Keywords: metabolic associated fatty liver disease; metabolic; nonalcoholic fatty liver disease (NAFLD); non-MR-NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5mL peripheral blood placed in sodium citrate vacuum tube, 5mL peripheral blood serum, 10mL random urine and 25g stool are collected at the baseline information and specimen collection. All these samples are used for screening potential indicators to evaluate prognosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic dysfunction-associated fatty liver disease (MAFLD) is a new concept proposed in 2020. Unlike non-alcoholic fatter liver disease (NAFLD), the diagnosis of MAFLD requires the presence any of the following 3 metabolic risks, including overweight/obesity, presence of diabetes mellitus, and evidence of metabolic dysregulation. However, there are patients that have hepatic steatosis but no metabolic risk, who thus do not meet the diagnostic criteria of MAFLD. Besides, there are patients with both MAFLD and other liver diseases. The clinical features and the management of these patients remain unclear. Thus, further histopathological and clinical study is required to elucidate and compare the characteristics of MAFLD and NAFLD.

Here, in this single-center, prospective clinical study, investigators are planning to establish a long-term follow-up cohort of patients with either MAFLD or NAFLD. In order to understand the risk of developing liver-related complications and important extra-hepatic outcomes (e.g. cardiovascular disease), and also to better elucidate the risk of disease progression in "lean" NAFLD individuals without any metabolic dysregulation and MAFLD individuals with dual or multiple causes.

Ultimately, investigators aim to improve the diagnosis of MAFLD and improve patients' outcomes.

DETAILED DESCRIPTION:
The study is divided into 2 parts:

Firstly, it contains a cross-sectional study to collect the clinical data of the patients with fatty liver. The clinical features of this population will be analysed.

Secondly, the study will collect the plasma, urine and stool samples of the patients in this cohort. And then a long-term follow-up of these patients will be carried out. Investigators wish to find out biomarkers that can detail patient stratification and predict the prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as hepatic steatosis in adults (fulfill at least one of the followings):

  1. Liver ultrasound shows liver parenchymal hyperechoic or "bright liver"
  2. Controlled attenuation-parameter (CAP) ≥248dB/m
  3. Hepatic steatosis diagnosed by CT/MRI/MRS
  4. MRI-based proton-density fat fraction (MRI-PDFF) shows liver fat content>8%
  5. Fatty liver confirmed by liver histology.

Exclusion Criteria:

1. Diagnosed with hepatocellular carcinoma or other malignancy (in accordance with the appropriate diagnostic criteria);
2. During pregnancy;
3. Patients with history of liver transplantation;
4. Patients with serious cardiovascular and cerebrovascular events (such as acute myocardial infarction, cerebral infarction, cerebral hemorrhage, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study include 3000 patients diagnosed as hepatic steatosis (both inpatients and outpatients of Nanfang hospital). We exclude the patients with history of liver transplantation, history of hepatocellular carcinoma (HCC) or other active malignancy, congestive heart failure and serious cerebrovascular disease, and pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2030-08-17 (Estimated); Study Completion 2030-08-17 (Estimated)

PRIMARY OUTCOMES:
All cause death | 10 years
  Noticed death of patient at follow-up visit

SECONDARY OUTCOMES:
Liver-related complications and important extra-hepatic outcomes (e.g. cardiovascular disease) | 10 years
  Noticed liver-related complications and important extra-hepatic outcomes (e.g. cardiovascular disease) of patient at follow-up visit
The correlation between different metabolic components and the clinical manifestations and disease progression | 10 years
  Risks of developing liver-related complications and important extra-hepatic outcomes

OTHER OUTCOMES:
The clinical manifestations and differences of metabolic-related fatty liver disease combine with different liver diseases | 10 years
  the clinical manifestations and long-term prognosis MAFLD with multiple or dual causes

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided